CLINICAL TRIAL: NCT00058617
Title: Administration of Neomycin Resistance Gene Marked EBV Specific Cytotoxic T-Lymphocytes to Patients With Relapsed EBV-Positive Lymphoma
Brief Title: Epstein Barr Virus (EBV) Specific Cytotoxic T-Cells, Relapsed Lymphoma, ANGEL
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: The Methodist Hospital Research Institute (Other); Center for Cell and Gene Therapy, Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Helen Heslop, Professor, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6423-ANGEL; ANGEL (Other: Baylor College of Medicine); NCT00002821 (obsolete NCT alias)
Record Dates: First submitted 2003-04-08; First posted 2003-04-09 (Estimated); Last update posted 2017-02-15 (Actual); Status verified 2017-02

CONDITIONS: Epstein-Barr Virus-Related Hodgkin Lymphoma; Epstein-Barr Virus-Related Non-Hodgkin Lymphoma; EBV Positive Plasma Cell Neoplasm
Keywords: EBV Positive Hodgkin's Lymphoma; EBV Positive Non-Hodgkin's Lymphoma; EBV Specific Cytotoxic T-Lymphocytes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Injection of EBV Specific CTLs (Experimental): Subjects will receive autologous EBV Specific CTLs. Patients that agree will recieve CTLs that have been marked with the neomycin resistance gene.
  Interventions: Biological: Injection of EBV Specific CTLs

INTERVENTIONS:
Biological: Injection of EBV Specific CTLs — Each patient will receive two injections, 14 days apart, according to the following dosing schedules:
  Group One Day 0 2x10^7 cells/m2 Day 14 2x10^7 cells/m2
  Group Two Day 0 2x10^7 cells/m2 Day 14 1x10^8 cells/m2
  Group Three Day 0 1x10^8 cells/m2 Day 14 2x 10^8 cells/m2
  If patients with active disease have stable disease or a partial response by the RECIST criteria at their 8 week or subsequent evaluations they are eligible to receive up to 6 additional doses of CTLs at monthly intervals-each of which will consist of the same cell number as their second injection. Patients will not be able to receive additional doses until the initial safety profile is completed at 6 weeks following the second infusion.

SUMMARY:
Patients have a type of lymph gland cancer called Hodgkin or non-Hodgkin Lymphoma which has come back or not gone away after treatment, including the best treatment known for relapsed Lymphoma.

Patients are being asked to volunteer to be in a research study using Epstein Barr virus specific cytotoxic T lymphocytes, a new experimental therapy. This therapy has never been used in patients with Hodgkin disease or this type of non-Hodgkin Lymphoma but it has been used successfully in children with other types of blood cancer caused by EBV after bone marrow transplantation. Some patients with Hodgkin or non-Hodgkin Lymphoma show evidence of infection with the virus that causes infectious mononucleosis Epstein Barr virus before or at the time of their diagnosis of the Lymphoma. EBV is often found in the cancer cells suggesting that it may play a role in causing Lymphoma. The cancer cells infected by EBV are very clever because they are able to hide from the body's immune system and escape destruction. Investigators want to see if it's possible to grow special white blood cells, called T cells, that have been trained to kill EBV infected cells.

Purpose The purpose of this study is to find the largest safe dose of EBV specific cytotoxic T cells, to learn what the side effects are and to see whether this therapy might help patients with Hodgkin disease and non-Hodgkin Lymphoma.

DETAILED DESCRIPTION:
The investigators will take 60-70 ml (12 teaspoonfuls) of blood from the patient to make a B cell line called a lymphoblastoid cell line or LCL by infecting the blood with a laboratory strain of EBV called B95-8. The investigators will then use this EBV infected cell line (which have been treated with radiation so that they cannot grow) as stimulator cells and mix it with more blood. This stimulation will train the T cells to kill EBV infected cells and result in the growth of an EBV specific T cell line. The investigators will then test the T cells to make sure that they kill the EBV infected cells and not normal cells and freeze them.

Patients will be entered into one of three different dosing schedules being evaluated. Three to six patients will be evaluated on each dosing schedule. Escalation will continue until irreversible or life threatening side effects considered to be related to the T cells are seen.

The cells will then be thawed and injected into the patients' vein over 10 minutes, after pretreatment with Tylenol and Benadryl. Tylenol and Benadryl are given to prevent a possible allergic reaction to the T cell administration. Initially, two doses of T cells will be given two weeks apart. If after the second infusion there is a reduction in the size of the patient's lymphoma on CT or MRI scan as assessed by a radiologist, the patient can receive up to six additional doses of the T cells. All of the treatments will be given at Texas Children's Hospital or the Methodist Hospital.

Patients will be followed in the clinic after the injections. To learn more about the way the T cells are working and how long they last in the body, an extra 40 mls (8 teaspoonfuls) of blood will be taken before each infusion and then 24 hours after each infusion, 3-4 days after each infusion and at 1, 2, 4, and 6 weeks post infusion and then at 3, 6, 9 and 12 months post infusion. The blood may be drawn from the central line at the time of regular blood tests. This blood will be used to test for the frequency and activity of EBV specific T cells. A total of at least 122 teaspoons (approximately 40 tablespoons) of blood will be collected during participation in this study.

If the patient decide to withdraw at any time during the study both samples and data collected during participation will be maintained.

ELIGIBILITY:
INCLUSION CRITERIA:

* Any patient with EBV positive Hodgkin disease or non-Hodgkin Lymphoma, or plasma cell neoplasms in second relapse regardless of age or sex, in first relapse or with primary disease or in first remission if immunosuppressive chemotherapy contraindicated, e.g. patients who develop Hodgkin disease after solid organ transplantation or if the Lymphoma is a second malignancy e.g. a Richters transformation of CLL.
* Life expectancy of greater than 6 weeks.
* No severe intercurrent infection
* Patient, parent/guardian able to give informed consent
* Bilirubin <2x normal,
* SGOT <3x normal,
* Hgb greater than 8.0 g/L
* Creatinine <2x normal for age
* Must have been off other investigational therapy for one month prior to entry in this study.
* Karnofsky score of greater than or equal to 50.

EXCLUSION CRITERIA:

* Patient with an EBV positive NHL secondary to an acquired immunodeficiency.
* Patients who are HIV positive
* Patient, parent/guardian unable to give informed consent
* Patients with a Karnofsky score of < 50.
* Patients with a life expectancy of <6 weeks
* Patients with a bilirubin greater than 2x normal. SGOT greater than 3x normal
* Patients with a creatinine greater than 2x normal for age
* Due to unknown effects of this therapy on a fetus, pregnant women are excluded from this research. The male partner should use a condom.

Note: Patients who would be excluded from the protocol strictly for laboratory abnormalities can be included at the investigator's discretion after approval by the CCGT Protocol Review Committee and the FDA reviewer.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 1996-01; Primary Completion 2011-08 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
The safety of two IV injections of auto EBV specific CTLs will be determined through adverse event measurement. These CTLs may be marked with the neomycin resistance gene introduced by a retroviral vector. | 6 weeks
  Three patients will be enrolled at the first dose level and followed for six weeks after the second dose (which will constitute a course) for evaluation of any critical toxicity. The toxicity will be evaluated as per the NCI Common Toxicity criteria version 2.0.Any toxicity scored as Grade 3 or 4 according to this criteria will be classified as an adverse event. If no toxicity is observed in the first three patients then we will enroll another three patients at the next dose level. However, if toxicity is observed in no more than one out of the three patients then three more patients will be enrolled at the same dose level. Now if the toxicity is observed in no more than one out of the six patients then we will advance to the next dose level and enroll three new patients. If toxicity is observed in two or more patients out of six then the dose limiting toxicity (DLT) has been exceeded and the previous dose level will be considered as the maximum tolerated dose (MTD) level.
To determine the feasibility of generating EBV specific cytotoxic T cell lines from patients with active EBV positive Lymphoma including Hodgkin Disease (HD) or Non-Hodgkin Lymphoma (NHL). | 6 weeks
To determine the survival, immunological efficacy and anti-tumor effects of EBV specific cytotoxic T-lymphocyte lines. | 15 years
  During the course of the study the survival, immunological efficacy and anti-tumor activity of neomycin resistance gene marked EBV specific cytotoxic T-lymphocyte lines will also be studied. In order to gain reasonable insight into the anti-tumor activity and late toxicity the patients will be followed for a total of twelve weeks.In the present case, the chances of observing any late toxicity should be if anything lower, as in this case the CTLs will be derived autologously.

CONTACTS AND LOCATIONS:
Overall Officials: Helen E Heslop, MD, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Houston Methodist Hospital, Houston, Texas
  - Texas Children's Hospital, Houston, Texas